CLINICAL TRIAL: NCT00789529
Title: Objective Testing of Tear Film Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manhattan Vision Associates (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CS-101
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-04

CONDITIONS: Contact Lens Solutions
Keywords: Contact lenses, wettability, Contact Lens Disinfectant Solutions, pre-lens tear film

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Opti-Free® RepleniSH® MPDS
  Interventions: Device: Opti-Free® RepleniSH® MPDS
- 2 (Active Comparator): Renu MultiPlus®
  Interventions: Device: ReNu MultiPlus®

INTERVENTIONS:
Device: Opti-Free® RepleniSH® MPDS — soft contact lens disinfecting solution
  Arms: 1
Device: ReNu MultiPlus® — soft contact lens disinfecting solution
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the in-vivo wettability of soft contact lenses when cared with two different multi-purpose solutions over a two week wearing period.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be at least 18 years of age and no more than 80 years of age.
2. The subject must have a best corrected visual acuity of 20/30 or better for each eye.
3. The subject must habitually wear contact lenses.
4. The subject must have had an eye exam within the last 12 months. The exam data must be available to the investigators prior to the first visit.
5. The subject must have normal eyes, no use of ocular medications, no ocular infection of any type, and no ocular inflammation.
6. The subject must read understand and sign the Statement of Informed Consent.
7. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

1. Ocular or systemic allergies or disease that might interfere with contact lens wear.
2. Systemic disease, autoimmune disease or use of medication which might interfere with contact lens wear.
3. Clinically significant (FDA Scale grade 3 or 4) corneal edema, corneal vascularization, corneal staining or any other abnormalities of the cornea which would contraindicate contact lens wear.
4. Clinically significant (FDA Scale grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
5. Any ocular infection.
6. Pregnancy or lactation.
7. Diabetes
8. Infectious diseases (e.g. hepatitis, tuberculosis)
9. Contagious immunosuppressive diseases (e.g. HIV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Zikos, OS, MS, Principal Investigator — MVA/IVR
Locations (1):
- MVA/IVR, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of patients was conducted by approaching the patients seen in the practice.
Pre-assignment Details: 32 subjects were recruited and enrolled in the study. No subjects had to be excluded.
Groups:
- 1 - ReNu MultiPlus First, Opti-Free RepleniSH Second: Used ReNu MultiPlus multi-purpose solution for the care of new contact lenses in the first intervention period, and used Opti-Free RepleniSH multi-purpose disinfecting solution for the care of new contact lenses in the second intervention period
- 2 - Opti-Free RepleniSH First, ReNu MultiPlus Second: Used Opti-Free RepleniSH multi-purpose disinfecting solution for the care of new contact lenses in the first intervention period, and used ReNu MultiPlus multi-purpose solution for the care of new contact lenses in the second intervention period
Period: Overall Study
Arm/Group | 1 - ReNu MultiPlus First, Opti-Free RepleniSH Second | 2 - Opti-Free RepleniSH First, ReNu MultiPlus Second
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other Reason | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 - ReNu MultiPlus First: Used ReNu MultiPlus first, Opti-Free RepleniSH Second
- 2 - Opti-Free RepleniSH First: Opti-Free RepleniSH first, ReNu MultiPlus Second
- Total: Total of all reporting groups
Arm/Group | 1 - ReNu MultiPlus First | 2 - Opti-Free RepleniSH First | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.3 (3.8) | 27.4 (5.1) | 27.3 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Objective, In-vivo Soft Contact Lens Wettability Index
Description: The wettability index is derived from the slope of a metric developed to measure the regularity of the Shack-Hartmann wavefront sensor image. The more wettable a lens is the more stable the metric and the slope of the metric (the wettability index) is closer to zero. The more negative values indicate a less wettable the lens.
Time Frame: 2 weeks
Population: Per protocol. All participants that completed both arms were analysed.
Measure: Mean (Standard Deviation); unit: wettability index
Groups:
- Opti-Free® RepleniSH® MPDS: Used Opti-Free® RepleniSH® MPDS
- Renu MultiPlus®: Used Renu MultiPlus®
Arm/Group | Opti-Free® RepleniSH® MPDS | Renu MultiPlus®
Number analyzed (Participants) | 30 | 30
wettability index | -1.82 (2.88) | -1.98 (2.80)

2. Secondary Outcome: Subject Questionnaire Response
Description: Subject questionnaire response: Overall comfort at 2 weeks in a 0-50 point scale.
  0=Very poor 50 = Excellent
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opti-Free® RepleniSH® MPDS | Renu MultiPlus®
Number analyzed (Participants) | 30 | 30
units on a scale | 42.7 (7.3) | 43.1 (5.0)

ADVERSE EVENTS:
Time Frame: Length of study was 24 to 32 days.
Arm/Group | 1 - ReNu MultiPlus First | 2 - Opti-Free RepleniSH First
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less